CLINICAL TRIAL: NCT07087821
Title: Economic Evaluation of Managing Epilepsy Well (MEW) Network Epilepsy Self-Management Programs
Brief Title: NYU Epilepsy Self-Management Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-00151; U48DP006844 (NIH)
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RCT 1: UPLIFT (Experimental): Participants in RCT 1 assigned to the UPLIFT arm.
  Interventions: Behavioral: UPLIFT
- RCT 1: Enhanced Usual Care (Active Comparator): Participants in RCT 1 assigned to the enhanced usual care arm.
  Interventions: Behavioral: Enhanced Usual Care
- RCT 2: PACES (Experimental): Participants in RCT 2 assigned to the PACES arm.
  Interventions: Behavioral: PACES
- RCT 2: Enhanced Usual Care (Active Comparator): Participants in RCT 2 assigned to the enhanced usual care arm.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: UPLIFT — UPLIFT is an 8-week epilepsy self-management programs delivered to small groups of people with epilepsy (PWE) by Webex. UPLIFT is focused on self-management of depressive symptoms.
  Each weekly session is 1 hour long and is comprised of a check-in period, teaching on the week's topic, group discussion, a skill-building exercise and a home practice assignment.
  Arms: RCT 1: UPLIFT
Behavioral: PACES — PACES is an 8-week epilepsy self-management programs delivered to small groups of people with epilepsy (PWE) by Webex. PACES focuses on general epilepsy self-management.
  Each weekly session is 1 hour long and is comprised of a check-in period, teaching on the week's topic, group discussion, a skill-building exercise and a home practice assignment.
  Arms: RCT 2: PACES
Behavioral: Enhanced Usual Care — Participants receive referrals to local epilepsy support groups.
  Arms: RCT 1: Enhanced Usual Care; RCT 2: Enhanced Usual Care

SUMMARY:
The investigators will conduct two-arm randomized controlled trials (RCTs) comparing effects of UPLIFT vs. enhanced usual care and PACES vs. enhanced usual care, respectively, on quality of life, depressive symptoms and seizures over 12 months in NYU patients with epilepsy.

DETAILED DESCRIPTION:
UPLIFT and PACES are two evidence-based epilepsy self-management programs whose adoption and impact are limited by the lack of sustainable funding models.

The investigators will conduct an economic evaluation of these programs using data from completed and new trials in both healthcare and community settings.

The investigators will conduct two parallel RCTs to compare effects of UPLIFT vs. enhanced usual care, and separately, PACES vs. enhanced usual care.

Outcome data including patient-reported outcomes and costs will be aligned across the two trials and community implementation and collected at baseline and 3-, 6-, and 12-month follow-up visits for use in the economic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* English-speaking (UPLIFT and PACES) or Spanish-speaking (UPLIFT only).
* Diagnosed with epilepsy for at least one year
* Able to understand the informed consent and provide consent
* Elevated depressive symptoms - Patient Health Questionnaire-9 (PHQ-9) score ≥10; applies to UPLIFT only

Exclusion Criteria:

* Severe depressive symptoms (score of ≥20 on PHQ-9)
* Active suicidal ideation (score of ≥1 on PHQ-9 item #9 or otherwise reported during screening)
* Active psychotic disorder (psychiatric diagnosis and/or antipsychotic medications in the electronic health records (EHR)
* Significant cognitive impairment (indicated in the EHR or evident during screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-18 (Estimated); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Patient Health Questionnaire-9 (PHQ-9) Score <5 | Baseline
  RCT 1 participants only.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression. The primary outcome is the count of participants who score less than 5 on the PHQ-9 (i.e., absence of clinically significant depressive symptoms).
Number of Participants with PHQ-9 Score <5 | Post-Intervention Month 3 Follow-up (Approximately Month 5)
  RCT 1 participants only.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression. The primary outcome is the count of participants who score less than 5 on the PHQ-9 (i.e., absence of clinically significant depressive symptoms).
Number of Participants with PHQ-9 Score <5 | Post-Intervention Month 6 Follow-up (Approximately Month 8)
  RCT 1 participants only.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression. The primary outcome is the count of participants who score less than 5 on the PHQ-9 (i.e., absence of clinically significant depressive symptoms).
Number of Participants with PHQ-9 Score <5 | Post-Intervention Month 12 Follow-up (Approximately Month 14)
  RCT 1 participants only.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression. The primary outcome is the count of participants who score less than 5 on the PHQ-9 (i.e., absence of clinically significant depressive symptoms).
Composite PHQ-9 and Quality of Life in Epilepsy Inventory-31 (QOLIE-31) Score | Baseline
  RCT 2 participants only.
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
  The scores from both the PHQ-9 and QOLIE-3 are re-scaled into a combined, Composite PHQ+QOLIE Score ranging from 0-100; higher values indicate more favorable outcomes.
Composite PHQ-9 and Quality of Life in Epilepsy Inventory-31 (QOLIE-31) Score | Post-Intervention Month 3 Follow-up (Approximately Month 5)
  RCT 2 participants only.
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
  The scores from both the PHQ-9 and QOLIE-3 are re-scaled into a combined, Composite PHQ+QOLIE Score ranging from 0-100; higher values indicate more favorable outcomes.
Composite PHQ-9 and QOLIE-31 Score | Post-Intervention Month 6 Follow-up (Approximately Month 8)
  RCT 2 participants only.
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
  The scores from both the PHQ-9 and QOLIE-3 are re-scaled into a combined, Composite PHQ+QOLIE Score ranging from 0-100; higher values indicate more favorable outcomes.
Composite PHQ-9 and QOLIE-31 Score | Post-Intervention Month 12 Follow-up (Approximately Month 14)
  RCT 2 participants only.
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
  The scores from both the PHQ-9 and QOLIE-3 are re-scaled into a combined, Composite PHQ+QOLIE Score ranging from 0-100; higher values indicate more favorable outcomes.
5-level EQ-5D version (EQ-5D-5L) Score | Baseline
  The EQ-5D-5L is a standardized questionnaire used to measure health-related quality of life (HRQoL). It consists of two parts: a descriptive system and a visual analogue scale (EQ VAS). The descriptive system assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. The EQ VAS provides a self-assessment of overall health on a scale of 0 to 100, where higher scores indicate better health. The EQ-5D-5L will be used to derive utility values to estimate quality-adjusted life years (QALYs) for cost-utility analyses.
EQ-5D-5L Score | Post-Intervention Month 3 Follow-up (Approximately Month 5)
  The EQ-5D-5L is a standardized questionnaire used to measure health-related quality of life (HRQoL). It consists of two parts: a descriptive system and a visual analogue scale (EQ VAS). The descriptive system assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. The EQ VAS provides a self-assessment of overall health on a scale of 0 to 100, where higher scores indicate better health. The EQ-5D-5L will be used to derive utility values to estimate quality-adjusted life years (QALYs) for cost-utility analyses.
EQ-5D-5L Score | Post-Intervention Month 6 Follow-up (Approximately Month 8)
  The EQ-5D-5L is a standardized questionnaire used to measure health-related quality of life (HRQoL). It consists of two parts: a descriptive system and a visual analogue scale (EQ VAS). The descriptive system assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. The EQ VAS provides a self-assessment of overall health on a scale of 0 to 100, where higher scores indicate better health. The EQ-5D-5L will be used to derive utility values to estimate quality-adjusted life years (QALYs) for cost-utility analyses.
EQ-5D-5L Score | Post-Intervention Month 12 Follow-up (Approximately Month 14)
  The EQ-5D-5L is a standardized questionnaire used to measure health-related quality of life (HRQoL). It consists of two parts: a descriptive system and a visual analogue scale (EQ VAS). The descriptive system assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. The EQ VAS provides a self-assessment of overall health on a scale of 0 to 100, where higher scores indicate better health. The EQ-5D-5L will be used to derive utility values to estimate quality-adjusted life years (QALYs) for cost-utility analyses.

SECONDARY OUTCOMES:
Change from Baseline in PHQ-9 Score | Baseline, Post-Intervention Month 3 Follow-up (Approximately Month 5)
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
Change from Baseline in PHQ-9 Score | Baseline, Post-Intervention Month 6 Follow-up (Approximately Month 8)
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
Change from Baseline in PHQ-9 Score | Baseline, Post-Intervention Month 12 Follow-up (Approximately Month 14)
  The PHQ-9 is a 9-item assessment of depression; each item is rated on a scale from 0-3. The total score is the sum of item responses and ranges from 0-27; higher scores indicate greater levels of depression.
Change from Baseline in QOLIE-31 | Baseline, Post-Intervention Month 3 Follow-up (Approximately Month 5)
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
Change from Baseline in QOLIE-31 | Baseline, Post-Intervention Month 6 Follow-up (Approximately Month 8)
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
Change from Baseline in QOLIE-31 | Baseline, Post-Intervention Month 12 Follow-up (Approximately Month 14)
  The QOLIE-31 is a 31-item questionnaire evaluating an epilepsy patient's quality of life (QOL) perception. The overall score is derived by weighing and then summing the 7 domain scores, which correspond with the item responses. The overall score is converted to a final, 0-100 point score, where higher converted scores reflect better QOL.
Change from Baseline in Seizure Frequency | Baseline, Post-Intervention Month 3 Follow-up (Approximately Month 5)
Change from Baseline in Seizure Frequency | Baseline, Post-Intervention Month 6 Follow-up (Approximately Month 8)
Change from Baseline in Seizure Frequency | Baseline, Post-Intervention Month 12 Follow-up (Approximately Month 14)
Healthcare Utilization | Baseline
  A composite count of outpatient visits, hospitalizations, and emergency department visits will be collected using a combination of EHR review and patient self-report.
Healthcare Utilization | Post-Intervention Month 3 Follow-up (Approximately Month 5)
  A composite count of outpatient visits, hospitalizations, and emergency department visits will be collected using a combination of EHR review and patient self-report.
Healthcare Utilization | Post-Intervention Month 6 Follow-up (Approximately Month 8)
  A composite count of outpatient visits, hospitalizations, and emergency department visits will be collected using a combination of EHR review and patient self-report.
Healthcare Utilization | Post-Intervention Month 12 Follow-up (Approximately Month 14)
  A composite count of outpatient visits, hospitalizations, and emergency department visits will be collected using a combination of EHR review and patient self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health - NYU Langone Hospital-Brooklyn, Brooklyn, New York
  - NYU Langone Health - NYU Comprehensive Epilepsy Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Tanya.Spruill@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to Tanya.Spruill@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.